CLINICAL TRIAL: NCT01309893
Title: A Study to Evaluate the Product Feasibility of a New Silicone Hydrogel Contact Lens
Brief Title: A Study to Evaluate a New Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 687E
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Myopia
Keywords: Contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Lens (Experimental): Bausch & Lomb investigational silicone hydrogel contact lens for 1 week; then issued Air Optix Aqua Lens for 1 week.
  Interventions: Device: Investigational Lens; Device: Air Optix Aqua lens
- Air Optix Aqua Lens (Active Comparator): Ciba Vision Air Optix Aqua contact lens for 1 week; then issued Investigational Lens for 1 week.
  Interventions: Device: Investigational Lens; Device: Air Optix Aqua lens

INTERVENTIONS:
Device: Investigational Lens — Lenses worn on a daily wear basis for one week
Device: Air Optix Aqua lens — Lenses worn on a daily wear basis for one week

SUMMARY:
The objective of this study is to determine the clinical feasibility and to evaluate the product performance of investigational contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* Be myopic and require lens correction from -0.50 D to -5.50 D in each eye.

Exclusion Criteria:

* Any systemic disease affecting ocular health.
* Using any systemic or topical medications that will affect ocular physiology or lens performance.
* An active ocular disease, any corneal infiltrative response or are using any ocular medications.
* Any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, OD, MS, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited for this 2-week study conducted at three investigational sites in the USA. The first participant was enrolled on 12/17/2010; the last participant exited the study on 01/20/2011.
Pre-assignment Details: 66 participants enrolled; 64 participants completed. Half wore Investigational Lens for 1 week then crossed over to Air Optix Aqua lens for 1 week. The other half wore Air Optix Aqua Lens for 1 week then crossed over to Investigational Lens for 1 week. The order of lens use was randomized and participant-masked.
Groups:
- Investigational Lens First, Then Air Optix Aqua Lens: Enrolled participants spent 1 week using Investigational Lens, and then crossed over to 1 week using Air Optix Aqua lens. The order of contact lens use was randomized and participant-masked.
- Air Optix Aqua Lens First, Then Investigational Lens: Enrolled participants spent 1 week using Air Optix Aqua Lens, and then crossed over to 1 week using Investigational Lens. The order of contact lens use was randomized and participant-masked.
Period: Week 1 - First Intervention
Arm/Group | Investigational Lens First, Then Air Optix Aqua Lens | Air Optix Aqua Lens First, Then Investigational Lens
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0
Period: Week 2 - Crossover Intervention
Arm/Group | Investigational Lens First, Then Air Optix Aqua Lens | Air Optix Aqua Lens First, Then Investigational Lens
Started | 33 | 33
Completed | 32 | 32
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Missed crossover visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: All eligible enrolled participants
Groups:
- Entire Study Population: All eligible enrolled participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Distance High Contrast logMAR Visual Acuity at 1 Week
Description: Mean difference in distance high contrast logMAR over all lens VAs (visual acuity) from Baseline and 1 Week
Time Frame: Baseline & 1 week
Population: All eligible, dispensed eyes
Measure: Least Squares Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Investigational Lens: Bausch & Lomb investigational silicone hydrogel contact lens
  Investigational Lens: Lenses worn on a daily wear basis for one week
- Air Optix Aqua Lens: Ciba Vision Air Optix Aqua contact lens
  Air Optix Aqua lens: Lenses worn on a daily wear basis for one week
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Number analyzed (Participants) | 66 | 66
Number analyzed (eyes) | 132 | 132
logMAR | -0.031 (0.069) | -0.015 (0.071)

2. Secondary Outcome: Slit Lamp Findings ≥ Grade 2
Description: Slit lamp findings are measured on a scale of 0-4, where 0=none, and 4=severe. The slit lamp exam is a routine procedure done to evaluate eye health and determine eligibility for clinical trial. It provides view of the different parts of the eye. During the exam, a doctor can look at the front parts of the eye, including the cornea, the lens, the iris and other parts of the anterior segment of the eye. Fluorescein dye may be used during a slit lamp examination to make it easier to detect inflammation, infections, or injured area on the cornea.
Time Frame: 1 week
Population: All dispensed eyes
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Number analyzed (Participants) | 65 | 63
Number analyzed (eyes) | 130 | 126
eyes | 0 | 0

3. Secondary Outcome: Overall Comfort
Description: Comfort measured by participant on a scale of 0-100 with 100 being the most favorable.
Time Frame: 1 week
Population: All eligible dispensed eyes
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Number analyzed (Participants) | 63 | 63
Number analyzed (eyes) | 126 | 126
units on a scale | 57.3 (27.8) | 80.8 (27.2)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Investigational Lens | Air Optix Aqua Lens
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other